CLINICAL TRIAL: NCT04166656
Title: Multicenter, Randomized, Phase III, Trial Assessing the Immunogenicity and Safety of Three Meningococcal B Vaccine Strategies Among Patients With Asplenia
Brief Title: Research Trial Assessing the Immunogenicity and Safety of Three Meningococcal B Vaccine Strategies Among Patients With Asplenia.
Acronym: SPLEMENGO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: EUCLID Clinical Trial Platform (Other); Recherche Clinique Paris Descartes Necker Cochin Sainte Anne (Other); CIC 1417 Cochin-Pasteur (Other); Innovative clinical research in vaccinologie (I-REIVAC) (Unknown); Institut Pasteur (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P170938J; 2019-000924-17 (EudraCT Number)
Record Dates: First submitted 2019-08-29; First posted 2019-11-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Splenectomy
Keywords: Meningococcal B vaccine; vaccine strategies; splenectomized individuals
MeSH Terms: interventions — MenB-FHbp vaccine; 4CMenB vaccine

STUDY DESIGN:
Masking Description: The trial will be open label. However, the assessment of the primary and secondary immunological endpoints will be carried out blind from the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A : Trumenba®: Standard vaccination (Other): Two doses of 0.5 ml each at one month intervals, followed by a third dose given at 6 months after the second dose.
  Interventions: Biological: Trumenba®
- Arm B:Bexsero®: standard vaccination regimen (Other): Two doses of 0.5 ml each at one month intervals
  Interventions: Biological: Bexsero®
- Arm C : Bexsero® Innovative vaccine strategy (Other): Two doses of 0.5 ml each at one month intervals, followed by a third dose given at 6 months after the second dose.
  Interventions: Biological: Bexsero®

INTERVENTIONS:
Biological: Trumenba® — Trumenba® (Pfizer): Suspension for intramuscular injection in 0.5 mL single-dose prefilled.
  Arms: Arm A : Trumenba®: Standard vaccination
Biological: Bexsero® — Bexsero® (GSK): available as a suspension for intramuscular injection in a prefilled syringe
  Arms: Arm B:Bexsero®: standard vaccination regimen; Arm C : Bexsero® Innovative vaccine strategy

SUMMARY:
The purpose of the study is to evaluate the immunological response and tolerance of 3 vaccine strategies against meningococcus B, a potentially fatal invasive infection.

DETAILED DESCRIPTION:
Currently, in France, no immunogenicity data on Meningococcal B vaccines, neither with Bexsero® nor with Trumenba®, are available in asplenic patients, population at high risk of infection.

As asplenic individuals (all causes) show less optimal immune response to conjugate meningococcal C vaccine compared to matched controls. [4], we hypothesize that a similar less optimal response may be expected for MenB vaccines among asplenic subjects. .

That is why, we proposed in this study to evaluate two reinforced strategies with 3 administrations (M0, M1, and M6) of Bexsero® or Trumenba ®. Moreover, the study will also allow exploring the persistence of the immune response in this population. Indeed, few data are available on this persistence in the general population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, >=18 to <=75 years old.
2. Asplenic patient (for at least 2 weeks) with Howell Jolly bodies visible on blood film
3. Splenectomy confirmed by consultation and/or hospitalization report or the ultrasound if it has been performed during the routine follow-up
4. Women of childbearing age must have an effective contraception during the first 9 months of the study.
5. Participants must give written consent prior to any trial procedure
6. Participants must be covered by social security regimen or equivalent.
7. Participants will be followed during the 4 years from the inclusion visit.

Exclusion Criteria:

1. History of meningococcal vaccination B.
2. History of anaphylaxis post vaccination.
3. Known allergy to any components (active substances or excipients) of both vaccines.
4. Patients who cannot stop antibiotics 3 days before blood collection.
5. Participants who have received any another vaccines within 4 weeks prior to immunization or who are planning to receive any vaccine within the first 7 months of the study (except the meningococcal ACWY vaccine, the anti-pneumococcal vaccine, the Haemophilus influenzae type B vaccine, the anti-Covid-19 vaccine), annual influenza vaccination which is permitted 2 weeks before and after each vaccination visit of the study and then allowed at any time during the study follow up).
6. Parenteral Ig within the 3 months prior to VS or planned during the study.
7. Chemotherapy agents within 6 months prior M0 or planning to take any during the study.
8. Steroids (> 10mg/day; > 14 days) within the month preceding M0 or planning to take any during the study.
9. Any pathology or condition that may impair the immune response, apart from splenectomy: immunosuppressive therapy in progress or in the 6 months prior to inclusion, hematopoietic stem cells allo / autograft, primary immunodeficiency, nephrotic syndrome, evolutive cancer, cirrhosis, known infection to HIV;
10. Thrombocytopenia or any coagulation disorder contra-indicating intramuscularly injections.
11. Pregnancy, breastfeeding or positive pregnancy test up to 7 months after inclusion.
12. Severe acute febrile illness within the week before inclusion.
13. Registration for any other clinical trial throughout the trial period except observational study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders defined as participants with seroconversion | One month after the completeness of three anti-meningococci B vaccine strategies (at M7 for all arms) in asplenic adults.
  Proportion of responders defined as participants with seroconversion (i.e. hSBA titer increases from <4 before vaccination to at least 4) or with hSBA titer showing a 4-fold increase (if hSBA titer was at least 4 before vaccination) one month after the completeness of three anti-meningococci B vaccine strategies (at M7 for all arms) in asplenic adults.

SECONDARY OUTCOMES:
Immunogenicity | one month after the completeness of each vaccine strategy
  Immunogenicity at M2/M7, i.e. one month after the completeness of each vaccine strategy:
  * Serum bactericidal antibody (hSBA) Geometric Mean Titer (GMT).
  * Proportion of responding participants using the conservative threshold of 8.
  * Proportion of participants achieving an hSBA titer equal to or greater than the lower limit of quantification of the assay.
Persistence of immunogenicity | At M12 M24, M36 and M48
  Persistence of immunogenicity at M12 M24, M36 and M48 for each vaccine strategy
  * Serum bactericidal antibody (hSBA), GMT.
  * Proportion of responding participants using the conservative threshold of 8.
  * Proportion of participants achieving an SBA titre equal to or greater than the lower limit of quantification of the assay.
Modeling of the determinants of immunogenicity | during the trial
  Modeling of the determinants of immunogenicity: reason for splenectomy, age, gender, immunosuppressive or immunomodulatory agent
Any event or serious adverse event | 7 days following each vaccination.
  Any event or serious adverse event during the trial possibly or not related to vaccine immunization.
safety and effectiveness | through study completion
  To assess safety and effectiveness of Bexsero® and Trumenba® in asplenic adults older than 65 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Odile LAUNAY, MD,PhD, Principal Investigator — CIC 1417 Clinical Center Investigation; MUHAMED-KHEIR TAHA, MD, PHD, Study Director — Institut Pasteur
Locations (1):
- I-REIVAC/CIC1417 Cochin Hospital, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Borrow R. Advances with vaccination against Neisseria meningitidis. Trop Med Int Health. 2012 Dec;17(12):1478-91. doi: 10.1111/j.1365-3156.2012.03085.x. Epub 2012 Sep 4. PMID 22947250
- [Background] Frosi G, Biolchi A, Lo Sapio M, Rigat F, Gilchrist S, Lucidarme J, Findlow J, Borrow R, Pizza M, Giuliani MM, Medini D. Bactericidal antibody against a representative epidemiological meningococcal serogroup B panel confirms that MATS underestimates 4CMenB vaccine strain coverage. Vaccine. 2013 Oct 9;31(43):4968-74. doi: 10.1016/j.vaccine.2013.08.006. Epub 2013 Aug 14. PMID 23954380
- [Background] Murphy E, Andrew L, Lee KL, Dilts DA, Nunez L, Fink PS, Ambrose K, Borrow R, Findlow J, Taha MK, Deghmane AE, Kriz P, Musilek M, Kalmusova J, Caugant DA, Alvestad T, Mayer LW, Sacchi CT, Wang X, Martin D, von Gottberg A, du Plessis M, Klugman KP, Anderson AS, Jansen KU, Zlotnick GW, Hoiseth SK. Sequence diversity of the factor H binding protein vaccine candidate in epidemiologically relevant strains of serogroup B Neisseria meningitidis. J Infect Dis. 2009 Aug 1;200(3):379-89. doi: 10.1086/600141. PMID 19534597
- [Background] Balmer P, Falconer M, McDonald P, Andrews N, Fuller E, Riley C, Kaczmarski E, Borrow R. Immune response to meningococcal serogroup C conjugate vaccine in asplenic individuals. Infect Immun. 2004 Jan;72(1):332-7. doi: 10.1128/IAI.72.1.332-337.2004. PMID 14688112
- [Background] 5. Hcsp. Avis du hcsp relatif à l'utilisation du vaccin bexsero® (novartis vaccines and diagnostics). 2013. (link:http://www.hcsp.fr/explore.cgi/telecharger?nomfichier=hcspa20131025_vaccmeningocoquebbexsero®.pdf.
- [Background] McQuaid F, Snape MD, John TM, Kelly S, Robinson H, Houlden J, Voysey M, Toneatto D, Kitte C, Dull PM, Pollard AJ. Persistence of bactericidal antibodies to 5 years of age after immunization with serogroup B meningococcal vaccines at 6, 8, 12 and 40 months of age. Pediatr Infect Dis J. 2014 Jul;33(7):760-6. doi: 10.1097/INF.0000000000000327. PMID 24722351
- [Background] Wasserstrom H, Bussel J, Lim LC, Cunningham-Rundles C. Memory B cells and pneumococcal antibody after splenectomy. J Immunol. 2008 Sep 1;181(5):3684-9. doi: 10.4049/jimmunol.181.5.3684. PMID 18714044
- [Background] Mori M, Morris SC, Orekhova T, Marinaro M, Giannini E, Finkelman FD. IL-4 promotes the migration of circulating B cells to the spleen and increases splenic B cell survival. J Immunol. 2000 Jun 1;164(11):5704-12. doi: 10.4049/jimmunol.164.11.5704. PMID 10820247
- [Background] Sullivan JL, Ochs HD, Schiffman G, Hammerschlag MR, Miser J, Vichinsky E, Wedgwood RJ. Immune response after splenectomy. Lancet. 1978 Jan 28;1(8057):178-81. doi: 10.1016/s0140-6736(78)90612-8. PMID 74605
- [Background] Goldschneider I, Gotschlich EC, Artenstein MS. Human immunity to the meningococcus. I. The role of humoral antibodies. J Exp Med. 1969 Jun 1;129(6):1307-26. doi: 10.1084/jem.129.6.1307. PMID 4977280